CLINICAL TRIAL: NCT00747331
Title: Fenoldopam Prophylaxis of Splanchnic Organs Underperfusion During Cardiopulmonary Bypass: a Randomized, Controlled Trial.
Brief Title: Fenoldopam and Splanchnic Perfusion During Cardiopulmonary Bypass
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Marco Ranucci, M.D., IRCCS Policlinico S.Donato
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FenoldopamCPB
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2009-04-13 (Estimated); Status verified 2009-04

CONDITIONS: Cardiac Complications; Cardiopulmonary Bypass
Keywords: Cardiopulmonary bypass; Lactic acidosis; Oxygen delivery; Acute renal failure; outcome; cardiac; surgery
MeSH Terms: conditions — Acidosis, Lactic; Acute Kidney Injury | interventions — Fenoldopam; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Fenoldopam mesilate
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fenoldopam mesilate — Continuous intravenous infusion at 0.1 mcg/kg/min starting immediately before CPB and ending after 12 hours from the end of the operation
  Other Names: Corlopam
  Arms: A
Drug: Placebo — Intravenous infusion (saline)
  Infused at the same rate (ml/h) as the experimental drug
  Other Names: Saline
  Arms: B

SUMMARY:
Cardiopulmonary bypass (CPB) for cardiac operations may be accompanied by different patterns of visceral underperfusion. This could result in clinical patterns of lactic acidosis but in the most severe cases there is the risk for mesenteric infarction (0.2% of the cases). Renal function as well may be impaired due to a low oxygen delivery, and acute renal failure occurs in 1-2% of cases.

Fenoldopam mesilate is a selective splanchnic vasodilator when used at a dose < 0.1 mcg/kg/min.

The experimental hypothesis of this randomized, controlled trial (RCT) is that the use of fenoldopam may determine a better visceral perfusion during CPB.

DETAILED DESCRIPTION:
Randomized placebo-controlled double blinded study. Patients undergoing complex cardiac operations will be randomly allocated to the study or the control group.

All the patients will receive the standard of care of our Institution. Adequacy of CPB perfusion will be assessed using oxygen delivery calculation, lactate production, SvO2.

ELIGIBILITY:
Inclusion Criteria:

* Complex, combined cardiac operation
* Predicted CPB duration > 90 minutes

Exclusion Criteria:

* Age < 18 years
* No written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Peak blood lactate levels during CPB | 3 hours

SECONDARY OUTCOMES:
Urine output during CPB | 3 hours
Peak blood lactate levels during the postoperative period | 48 hours after the end of the operation
Peak serum creatinine level during the postoperative period | 48 hours after the end of the operation

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ranucci, M.D., Study Director — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico S.Donato, San Donato Milanese, Milan, Italy

REFERENCES:
- [Background] Ranucci M, Soro G, Barzaghi N, Locatelli A, Giordano G, Vavassori A, Manzato A, Melchiorri C, Bove T, Juliano G, Uslenghi MF. Fenoldopam prophylaxis of postoperative acute renal failure in high-risk cardiac surgery patients. Ann Thorac Surg. 2004 Oct;78(4):1332-7; discussion 1337-8. doi: 10.1016/j.athoracsur.2004.02.065. PMID 15464494
- [Derived] Esezobor CI, Bhatt GC, Effa EE, Hodson EM. Fenoldopam for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD012905. doi: 10.1002/14651858.CD012905.pub2. PMID 39607014
- [Derived] Ranucci M, De Benedetti D, Bianchini C, Castelvecchio S, Ballotta A, Frigiola A, Menicanti L. Effects of fenoldopam infusion in complex cardiac surgical operations: a prospective, randomized, double-blind, placebo-controlled study. Minerva Anestesiol. 2010 Apr;76(4):249-59. PMID 20332738